CLINICAL TRIAL: NCT00310557
Title: Multicenter, Open-label Study of the Safety (Open-label) and Efficacy (Open-label and Blinded Reader) of a Single Administration of Approximately 0.1 mmol/kg of Magnevist® Injection-enhanced Magnetic Resonance Arteriography (MRA) and 2-dimensional-time-of-flight (2D-TOF) MRA in Patients With Known or Suspected Renal Artery Disease Undergoing MRA of the Renal Arteries With Intra-arterial Digital Subtraction Arteriography (i.a. DSA) as the Standard of Reference
Brief Title: Magnevist® Injection-enhanced MRA Compared to Non Contrast MRA for the Detection of Stenosis of the Renal Arteries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 90940; 304629
Record Dates: First submitted 2006-03-31; First posted 2006-04-04 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Renal Artery Stenosis
MeSH Terms: conditions — Renal Artery Obstruction | interventions — Gadolinium DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Gadopentetate dimeglumine (Magnevist)

INTERVENTIONS:
Drug: Gadopentetate dimeglumine (Magnevist) — Approximately 0.1mmol/kg body weight, single intravenous administration on the study day

SUMMARY:
The purpose of this study is to look at the safety (what are the side effects) and efficacy (how well does it work) of Magnevist (the study drug) used for MRI of the renal arteries. The results will be compared to the results of MRI taken without Magnevist and with the results of your X-ray angiography.

DETAILED DESCRIPTION:
This study has previously been posted by Berlex, Inc. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc.Bayer HealthCare Pharmaceuticals, Inc.is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria: - Has known or suspected renal artery disease - Is scheduled for X-ray angiography Exclusion Criteria: - Has any contraindication to magnetic resonance imaging - Is scheduled for any procedure before the X-ray angiography - Had previously had stents placed bilaterally in the region to be imaged

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2003-12; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Accuracy, sensitivity and specificity based on quantitative assessment of stenosis | Image creation after injection - evaluation at blind read

SECONDARY OUTCOMES:
Diagnostic confidence | At blinded and/or open label read of images
Accuracy, sensitivity, and specificity based on visual assessment of stenosis assesses | At blinded and/or open label read of images
Difference in degree of stenosis | At blinded and/or open label read of images
Other diagnostic findings | At blinded and/or open label read of images
Localisation matching of maximum stenosis | At blinded and/or open label read of images
Image quality | At blinded and/or open label read of images
Image evaluability and presence of artifacts | At blinded and/or open label read of images
Proportions of correctly categorised arteries with regard to maximum stenosis | At blinded and/or open label read of images
Number of evaluable arteries | At blinded and/or open label read of images
Patient management | From baseline to 24 hours follow-up
Safety | From baseline to 24 hours follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer